CLINICAL TRIAL: NCT05683626
Title: Safety and Efficacy of Adalimumab Therapy for Treatment of Behcet's Disease-related Uveitis in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mervat Zidan Mahmoud, assistant lecturer, Sohag University
Other Study IDs: MZMahmoud
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Humira — subcutaneous injection

SUMMARY:
the goal of this prospective cohort study is to asses the Safety and efficacy of Adalimumab therapy for treatment of Behcet's disease-related uveitis in adult patients at sohag university hospital.

Patients will receive adalimumab (40 IU), subcutaneous injection every two weeks for 6 months either as a primary treatment or if refractory to corticosteroids and at least one conventional synthetic immunosuppressive drug.

DETAILED DESCRIPTION:
Study design: Prospective cohort study. Sample size: 40 eyes of adult patients with complete Behçet's disease associated uveitis either male or female will be included in the study.

1. Inclusion Criteria:

   Adult patients with complete Behçet's disease associated uveitis . BD was diagnosed according to the classification criteria for BD proposed by the International Study Group for Behçet Disease .
2. Exclusion Criteria:

   Any patient with HIV, HBV, HCV, syphilis, toxoplasma, tuberculosis or other infections; liver, renal, cardiac or demyelinating diseases as well as substance abuse and malignancies will be excluded from the study
3. Treatment plan:

Patients will receive adalimumab (40 IU), subcutaneous injection every two weeks for 6 months either as a primary treatment or if refractory to corticosteroids and at least one conventional synthetic immunosuppressive drug.

Patients will start adose of systemic corticosteroids (methylprednisolone 1mg/kg/day) ,it will be tapered based on clinical improvement of uveitis and systemic symptoms of behcet disease.

Also In case of anterior uveitis, topical prednisolone acetate 1% every hour and topical cyclopentolate hydrochloride 1% two or five times per day were prescribed. If it was necessary, pulse corticosteroid therapy was used (1 g/day, for 3-5 days) for severe uveitic attacks.

Evaluation:

All patients will be evaluated by a safety monitoring board including both ophthalmologist and a rheumatolgist who will be acknowledge in the acknowledgment section later on.

Follow up schedule ; 1st month, 3rd month and 6th month or in case of necessity (relapse or safety concerns).

Full ophthalmological examination will be done for all patients include;

1. slit lamp biomicroscopy.
2. VA testing (uncorrected and best corrected visual acuity)
3. intraocular pressure measurement.
4. fundus examination..
5. ocular coherence tomography.
6. flourescene angiography. Clinical data regarding BCVA, anterior chamber cells and vitreous cells will be collected at baseline ,3 month and at the end of follow-up; OCT will be performed at the start of therapy, at 3- and 6-month follow-up visit and whenever an ocular flare will be suspected.

FA will be performed at the start of therapy and at the end of follow up period.

The diagnosis of macular edema and vasculitis will be based on clinical, OCT, and angiographic findings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with complete Behçet's disease associated uveitis .

Exclusion Criteria:

* Any patient with HIV, HBV, HCV, syphilis, toxoplasma, tuberculosis or other infections; liver, renal, cardiac or demyelinating diseases as well as substance abuse and malignancies will be excluded from the study

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: 40 eyes of adult patients with complete Behçet's disease associated uveitis either male or female will be included in the study.
  Patients will receive adalimumab (40 IU), subcutaneous injection every two weeks for 6 months either as a primary treatment or if refractory to corticosteroids and at least one conventional synthetic immunosuppressive drug.
  Patients will start adose of systemic corticosteroids (methylprednisolone 1mg/kg/day) ,it will be tapered based on clinical improvement of uveitis and systemic symptoms of behcet disease.
  Also In case of anterior uveitis, topical prednisolone acetate 1% every hour and topical cyclopentolate hydrochloride 1% two or five times per day were prescribed. If it was necessary, pulse corticosteroid therapy was used (1 g/day, for 3-5 days) for severe uveitic attacks.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
BCVA | 1 year
  best corrected visual acuity

SECONDARY OUTCOMES:
AC cells | 1 year
  anterior chamber cells
vitreous haze | 1 year
  vitreous haze

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt